CLINICAL TRIAL: NCT03902483
Title: Role of Renal Doppler Ultrasound in Early Detection of Acute Kidney Injury in Critically Ill Patients
Brief Title: Renal Doppler Ultrasound in Early Detection of Acute Kidney Injury in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MANAR SALAH AHMED BARAKAT, Assiut University, Assiut University
Other Study IDs: MSA
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: renal doppler ultrasound — renal doppler ultrasound measuring renal resistive index

SUMMARY:
Acute kidney injury is a common complication of critical illness and is associated with high morbidity and mortality .Acute kidney injury is a syndrome that is characterized by a rapid decline in renal function and urine output, resulting in retention of waste products such as urea, nitrogen, and serum creatinine. Life-threatening consequences include volume overload, hyperkalaemia, and metabolic acidosis . In its severe form, Acute kidney injury requires renal replacement therapy, which is applied in 5±13% of Intensive Care Unit patients

DETAILED DESCRIPTION:
The incidence of Acute kidney injury in intensive care unit patients is rising due to the population age increasing, more comorbidities, and a higher prevalence of risk factors. Improved Intensive Care Unit management has, however, significantly diminished morbidity and the mortality of patients who develop Acute kidney injury I. Despite an increase in the number and severity of comorbidities, in-hospital mortality has declined, but the incidence of Acute kidney injury ,and Acute kidney injury requiring renal replacement therapy has increased over time .

There is still some dispute over the characterization of the different types of Acute kidney injury. Classically there are three types of Acute kidney injury: pre-renal, intrinsic renal, and post-renal failure. These are characterized as decreased renal blood flow (in 40-70% of the patients), direct (intrinsic) renal parenchymal damage (in 10-50% of the patients), and obstruction of urine flow which is less common in the ICU (10%), respectively..

In critically ill patients, sepsis and acute kidney injury are very common diseases and are associated with increased hospitalization and elevated in-hospital mortality rates Acute kidney injury is a dynamic process that evolves from an early reversible condition to an established disease and leads to sustained renal impairment, cell death ,and delayed renal recovery .Consequently, prompt resuscitation of the circulation and optimal perfusion pressure are the primary therapies for critically ill patients with Acute kidney injury. These methods are based principally on the appropriate management of intravenous fluid replacement and vasopressor administration under strict hemodynamic monitoring .

Mechanisms of Acute kidney injury comprise renal hypo-perfusion, intra-renal vasoconstriction, inflammation,oxidative stress and nephrotoxicity .An important pathophysiological pathway includes intra renal vasoconstriction and endothelial damage of the microvessels, leading to impaired macro- and microvascular flow, which further aggravates ischemia .

Renal vasoconstriction is an early manifestation of Acute kidney injury. More specifically, ultrasound imaging of the renal arteries can be instrumental in the early detection of Acute kidney injury. Indeed, renal blood flow is decreased at a nearly stage during acute tubular necrosis as a consequence of protracted intra renal vasoconstriction. The renal resistive index , which is used for assessing arterial pulsatility, was shown to correlate with renal vascular resistance . Renal Doppler ultrasound can measure the renal resistive index , a sonographic index that reflects alterations in blood flow profile of the intrarenal arcuate or interlobar arteries. It reflects the relation between the decline in speed loss of flow (flow velocity) between the peak of systole and the end of diastole in (renal) blood vessels: RRI = (peak systolic velocity _end diastolic velocity)/(peak systolic velocity). Normal values are reported between 0.60 and 0.70 with the difference between both kidneys mostly being less than 5% .

The Doppler renal resistive index has been used for years in a variety of clinical settings . Doppler imaging identifies changes in blood flow at the micro-vascular level. Evaluation of the vascular impedance at different sites of the renal parenchyma could provide useful diagnostic and prognostic information. An increase in renal vascular resistance may be an early sensitive sign of hemodynamic deterioration, even in seemingly stable patients.

Measuring flow resistance in the renal circulation, Renal resistive Index (RRI), could become part of vital organ function assessment using Doppler ultrasound. An increased Doppler Renal resistive Index is suggested to not only reflect changes in intra renal perfusion, but also in systemic hemodynamics .

Renal resistive index (RI), determined by Doppler ultrasonography, directly reveals and quantifies modifications in renal vascular resistance .

Aim of the work

The aim is to

1. Determine if the resistive Renal Index on ICU admission patients predicts the development of Acute kidney injury during the first week.
2. Determine whether resistive Renal Index is related to the severity of Acute kidney injury or not.

Patients and Methods 80 patients of critically ill patients including acute ischaemic insults, patients presenting with septicaemia, hypertension, respiratory failure, coagulation/ haemorrhagic disorders, shock, and liver disease and shock.

This study will be performed in the 24-bed mixed medical and surgical intensive care unit of the Assiut University Hospital.

Sample size calculations will be based on the assumption that patients not developing Acute kidney injury would have an RRI of 0.72 and patients developing Acute kidney injury would have an Acute kidney injury of 0.79 with a standard deviation of 0.11. These calculations were based on the results of other previous studies that reported median values for Acute kidney injury and no Acute kidney injury

AKI was defined according to the Kidney Disease Improving Global Outcome (KDIGO) classification using both creatinine and urine output criteria [20] KDIGO takes changes in creatinine within 48 hours, or a decline in the glomerular filtration rate (GFR) over 7 days, into account. AKI is defined as an increase in sCreat ≥0.3 mg/dL within 48 hours, or an increase in sCreat ≥1.5-times baseline, which is known or presumed to have occurred within the prior 7 days, or a Urine Out put of <0.5 mL/kg/h for 6 hours

Laboratory tests:

1. Complete blood count
2. Kidney function
3. Electrolytes including sodium,potassium, calcium,Phosphorus and uric acid
4. Urine analysis 5-24 hrs sodium in urine

Radiological test:

Doppler of both renal arteries with abdominal ultrasound. Renal resistive index was measured with ultrasound-Doppler

ELIGIBILITY:
Inclusion Criteria:

age >18 years ICU admission within 24 hours

Exclusion Criteria:

1. Poor abdominal echogenicity
2. Severe acute or chronic renal insufficiency
3. Dialysis dependency, renal transplantation
4. Renal artery stenosis, congenital renal diseases ,renal tumor
5. Suicidal attempt
6. Pregnancy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 80 patients of critically ill patients including acute ischaemic insults, patients presenting with septicaemia, hypertension, respiratory failure, coagulation/ haemorrhagic disorders, shock, and liver diseasea and shock.
  This study will be performed in the 24-bed mixed medical and surgical intensive care unit of the Assiut University Hospital.
  Sample size calculations will be based on the assumption that patients not developing Acute Kidney Injury would have an RRI of 0.72 and patients developing Acute Kidney Injury would have an Acute Kidney Injury of 0.79 with a standard deviation of 0.11. These calculations were based on the results of other previous studies that reported median values for Acute Kidney Injury and no Acute Kidney Injury
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Role of Doppler Renal resistative index in early Prediction of acute kidney injury in critically ill patients | at one day of the study
  Renal resistive index was measured with ultrasound-Doppler using atransparietal 5MHz pulsed-wave Doppler probe. After visualizing the kidney in ultrasound mode and checking for renal abnormalities, an arcuate or interlobar artery will be localized and three successive Doppler measurements at different positions in the kidney (high, middle and low) will be performed, 3 times in each kidney. So a total number of 9 RRI values will be obtained in each kidney.The median value of each section will be used and the 3 median values of each kidney will be averaged. patients developing AKI would have an AKI of 0.79 with a standard deviation of 0.11

CONTACTS AND LOCATIONS:
Overall Officials: abdalla ismael, Study Director — Dr.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellomo R, Kellum JA, Ronco C. Acute kidney injury. Lancet. 2012 Aug 25;380(9843):756-66. doi: 10.1016/S0140-6736(11)61454-2. Epub 2012 May 21. PMID 22617274
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Hilton R. Acute renal failure. BMJ. 2006 Oct 14;333(7572):786-90. doi: 10.1136/bmj.38975.657639.AE. No abstract available. PMID 17038736
- [Background] Basile DP, Anderson MD, Sutton TA. Pathophysiology of acute kidney injury. Compr Physiol. 2012 Apr;2(2):1303-53. doi: 10.1002/cphy.c110041. PMID 23798302
- [Background] Gomez H, Ince C, De Backer D, Pickkers P, Payen D, Hotchkiss J, Kellum JA. A unified theory of sepsis-induced acute kidney injury: inflammation, microcirculatory dysfunction, bioenergetics, and the tubular cell adaptation to injury. Shock. 2014 Jan;41(1):3-11. doi: 10.1097/SHK.0000000000000052. PMID 24346647
- [Background] Spatola L, Andrulli S. Doppler ultrasound in kidney diseases: a key parameter in clinical long-term follow-up. J Ultrasound. 2016 Apr 16;19(4):243-250. doi: 10.1007/s40477-016-0201-x. eCollection 2016 Dec. PMID 27965714
- [Background] Leoncini G, Martinoli C, Viazzi F, Ravera M, Parodi D, Ratto E, Vettoretti S, Tomolillo C, Derchi LE, Deferrari G, Pontremoli R. Changes in renal resistive index and urinary albumin excretion in hypertensive patients under long-term treatment with lisinopril or nifedipine GITS. Nephron. 2002 Feb;90(2):169-73. doi: 10.1159/000049038. PMID 11818701